CLINICAL TRIAL: NCT03114241
Title: Long-term Effects of a 3-month Pedometer-based Program to Enhance Physical Activity in Patients With Severe COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Basec-Nr. 2016-00151
Record Dates: First submitted 2017-03-22; First posted 2017-04-14 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COPD
Keywords: COPD; Physical activity; Endothelial function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to one of the two groups: conventional care group or intervention group. No minimization procedures are used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): An increase in step count of 15% compared to baseline will be set as the minimal goal for each patient during 3 months.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Intervention — Patients allocated to the intervention group receive a pedometer. They are encouraged to be more active by using the pedometer to measure the number of steps walked daily. An increase in step count of 15% compared to baseline will be set as the minimal goal for each patient. Monthly telephone calls are indicated to encourage compliance with the protocol and motivate patients to enhance their level of activity. The coached program ends after three months but patients keep their pedometer and are encouraged to sustain an increased level of daily physical activity for additional 9 months (end of study).
  Arms: Intervention

SUMMARY:
Long-term evaluation of a coaching program which helps patients with severe COPD to increase their daily step count, in addition to usual care.

DETAILED DESCRIPTION:
Daily physical activity (PA) is a predictor of survival in the general population and has become a significant outcome measure in patients with COPD. Recent studies have demonstrated an independent association between PA, hospitalizations and mortality. Increased PA has significant benefits for patients with COPD. In most studies PA has only been assessed at one time point. Little is known about longitudinal changes in PA and data on determinants of changes in PA are scant. Moreover, information on best approaches to enhance PA in a population with decreasing PA is missing. To evaluate the long-term effect of a coaching program which is aimed at helping patients with severe COPD (FEV1<50%) to enhance their level of daily physical activity, in addition to usual care. Furthermore, this study aims to evaluate mechanisms that are responsible for changes of physical activity over time such as sociodemographic factors, lung function, comorbidities, vascular function, exacerbations, and medication.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age ≥ 40 years
* Severe COPD (FEV1<50%) diagnosed according to GOLD-guidelines (www.goldcopd.org)

Exclusion Criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Acute or recent (within the last 6 weeks) exacerbation of COPD
* Attending a pulmonary rehabilitation program within the last 6 months
* Pregnant patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Difference between the changes in number of steps per day (assessed over one week) from baseline to 12 months in the intervention group compared to controls. | 12 months
  At visits, the number of steps per day will be assessed by a multisensory band (SenseWear Pro™; Bodymedia Inc., Pittsburgh, PA, USA) which will be worn on the upper left arm for 7 consecutive days.

SECONDARY OUTCOMES:
Assessment of endothelial function by flow-mediated dilatation | 12 months
  Flow-mediated dilatation measurements will be performed by ultrasonography of the brachial artery with a high-frequency (10.0-MHz) ultrasound-scanning probe proximal to the antecubital fossa. Flow mediated dilatation will be assessed by percent of baseline Diameter.

OTHER OUTCOMES:
Number of COPD exacerbations | 12 months
  The number of COPD exacerbations in the previous year and during the study period will be assessed
Height | 12 months
  Body height (meter)
Weight | months
  Body weight (Kilogram)
Blood pressure | 12 months
  Blood pressure (mmHg) is measured in triplicate separated by 1-minute intervals after resting in supine position for 5 minutes in a quiet room with a validated, semi-automated oscillometric device
Herat rate | 12 months
  Heart rate (bpm) is measured in triplicate separated by 1-minute intervals after resting in supine position for 5 minutes in a quiet room.
Blood gas analysis | 12 months
  Daytime blood gas analysis will be performed without supplemental oxygen and immediately analysed with a commercially available blood gas analyser (ABL90 Radiometer Copenhagen. Arterial pressure of oxygen (PaO2) and carbon dioxide (PaCO2) will be assessed. Further, oxygen saturation (SaO2) will be determined.
Questionnaire: Hospital Anxiety and Depression Scale (HADS): | 12 months
  The questionnaire is especially designed for patients with physical impairment and assesses their symptoms of anxiety and depression. There are 7 items for each domain (anxiety and depression). Agreement on statements is expressed on a scale from 0 to 3 and domain scores are calculated by summing up the scores for the 7 items resulting in scores from 0 (no anxiety/depression) to 21 (depression/anxiety very likely).
Questionnaire: COPD Assessment Test (CAT) | 12 months
  The test is designed to measure the impact of COPD on the patients' life and how this changes over time. The test includes 8 questions each with a scale from 0 to 5. The eight questions not only address respiratory or chest-related symptoms such as cough or sensation of mucus accumulation or chest tightness, but also more general complaints such as disturbances in sleep or decreased energy levels and daily limitations resulting from the disease. The total score will be assessed.
Questionnaire: Physical acitivity questionnaire | 12 months
  The questionnaire includes items about household activities, sport, and leisure time activities. The time and intensity spent at different physical acitivty levels will be assessed.
Questionnaire: Short-Form 36 (SF-36) Questionnaire | 12 months
  The SF-36 consists of eight scaled scores that are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The categories are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health
Comorbidities | 12 months
  The number and type of medical comorbidities will be assessed by interview.

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Clarenbach, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kohlbrenner D, Sievi NA, Senn O, Kohler M, Clarenbach CF. Long-Term Effects of Pedometer-Based Physical Activity Coaching in Severe COPD: A Randomized Controlled Trial. Int J Chron Obstruct Pulmon Dis. 2020 Nov 6;15:2837-2846. doi: 10.2147/COPD.S279293. eCollection 2020. PMID 33192057